CLINICAL TRIAL: NCT04763551
Title: Medically Assisted Procreation and Choice of the Embryo: How Far Would French People Like to go - An Opinion Survey Among Patients Resorting to in Vitro Fertilization (IVF) in France.
Brief Title: Medically Assisted Procreation and Choice of the Embryo: How Far Would French People Like to go
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0088
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Infertility
Keywords: Couple infertility with IVF indication; Genetic indication for PGD in France
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In today's context of bioethics laws revision concerning Medically Assisted Procreation, the investigators focus on the opinion of couples resorting to In Vitro Fertilization on a fundamental, much debated issue ; the choice of the embryo.

French lawmakers fear the investigators might be drifting towards embryo selection procedures, but no study allows us to state this is what patients request. This study aims at determining, among the population of patients who resort to Medically Assisted Procreation in France, the ratio of patients who are willing to select the embryo due to its genetic characteristics.

ELIGIBILITY:
Inclusion criteria:

- Male and female IVF patients in the MAP

Exclusion criteria:

- Patient not fluent in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female IVF patients in the MAP centers of Montpellier University Hospital, Jeanne de Flandres in Lille, and Foch Hospital in Paris (on request)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Medically Assisted Procreation | 1 day
  Determine, among the population of patients who resort to Medically Assisted Procreation in France, the ratio of patients who are willing to select the embryo due to its genetic characteristics

SECONDARY OUTCOMES:
Determine the type of embryo genetic selection | 1 day
  Determine the type of embryo genetic selection those patients request
Determine, among the population of patients who resort to Medically Assisted Procreation in France | 1 day
  Determine, among the population of patients who resort to Medically Assisted Procreation in France, the ratio of patients who are willing to select the embryo due to its genetic characteristics, according to the type of MAP (classical MAP, with or without gamete donation, MAP with PGD)

CONTACTS AND LOCATIONS:
Overall Officials: Noémie Ranisavljevic, M.D., Ph.D, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC